CLINICAL TRIAL: NCT03584347
Title: Evaluation of Physician Volumetric Accuracy During Hyaluronic Acid Soft Tissue Filler Injections and the Effect of Products' Biophysical Properties on an Injector's Performance: An Observational, Proof-of-concept Study
Brief Title: Evaluation of Physician Volumetric Accuracy During Filler Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erevna Innovations Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018-06-001
Record Dates: First submitted 2018-06-07; First posted 2018-07-12 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Injection Site

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Injection of filler material — Subjects will be blind folded and asked to deposit 0.2cc's of each of the four investigational products, in a randomized order. First, over a weight and then into a porcine membrane.

SUMMARY:
Objectives

1. Evaluate the ability of aesthetic physicians to accurately inject a specific amount (i.e., 0.2cc) of HA soft tissue filler; and
2. Investigate the effect of different HA gel properties (e.g., G', cohesivity, viscoelasticity) on an injector's performance accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Board-certified plastic surgeon, dermatologist, or oculoplastic surgeon.

Exclusion Criteria:

* N/A

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-06-03 (Actual); Primary Completion 2018-06-10 (Actual); Study Completion 2018-09-03 (Actual)

PRIMARY OUTCOMES:
Volumetric accuracy of HA filler injections using observational methods | Baseline
  physicians will attempt to inject 0.2CC of four HA products into a porcine membrane. Volumes will be measured in CC's and their accuracy assessed based on the amount of product left in the syringe.
Volumetric accuracy of HA filler expulsions over a scale | Baseline
  Physicians will attempt to dispense 0.2CC of four different HA products. They will do this into free air, over a scale. The weights will be calculated in grams and converted to CC's. The scale is the "Smart Weight" digital milligram scale, JDS20 edition. It's specifications are as follows: capacity: 20g/100ct/308.8gn/12.86dwt; readability: 0.001g/0.005ct/0.02gn/0.001dwt; scale dimensions: 3x5x0.8"; accuracy of 0.001grams and capacity of 20grams.

CONTACTS AND LOCATIONS:
Locations (1):
- Victoria Park Medispa, Westmount, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No